CLINICAL TRIAL: NCT02415998
Title: Transesophageal Echocardiography (TEE) to Guide and Confirm Epidural Catheters in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Kenichi Ueda (Other)
Responsible Party: Sponsor-Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201207769
Record Dates: First submitted 2015-04-06; First posted 2015-04-14 (Estimated); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Epidural Space
Keywords: TEE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TEE
  Interventions: Procedure: TEE

INTERVENTIONS:
Procedure: TEE — Epidural catheter will be placed under guidance of transesophageal echography in specific thoracic spinal segment.

SUMMARY:
The aim of this study is to assess whether transesophageal echocardiography (TEE) can be used to successfully guide an epidural catheter to a targeted thoracic level in pediatric patients. The catheter will be placed in the epidural space under real-time TEE imaging and assistance by a trained TEE operator (this could include an anesthesiologist or cardiologist).

DETAILED DESCRIPTION:
The aim of this study is to assess whether transesophageal echocardiography (TEE) can be used to successfully guide an epidural catheter to a targeted thoracic level in pediatric patients. The catheter will be placed in the epidural space under real-time TEE imaging and assistance by a trained TEE operator.

The primary outcome is to determine the success rate achieved using TEE guidance to thread an epidural catheter to a targeted thoracic spinal level. Post-operative radiograph will be used to confirm catheter position.

The secondary outcomes include analysis of catheter tip position within the epidural space as anterior, lateral or inferior to the spinal cord. Further, efficacy of the catheter will be determined using the following criteria from previous studies: Hemodynamic response at skin incision analyzed by heart rate and systemic blood pressure changes using the no change in HR or BP or changes < 20% from baseline were considered "sufficient block" to surgical stimulation, while HR or BP changes > 20% from baseline were considered "not sufficient block" to surgical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients scheduled to undergo cardiothoracic surgery or interventional cardiology diagnostic procedures under general anesthesia. All subjects will also be scheduled to undergo post-operative chest x-ray as a routine part of their clinical care, so no additional exposure to ionizing radiation will occur due to this study.

Exclusion Criteria:

* patients with known esophageal abnormalities, lesions or disease that would disqualify the patient for the use of TEE as standard procedure. We will further exclude any patients that are solely undergoing TEE diagnostic procedures and only include patients that are already scheduled to undergo procedures where TEE is used as part of routine surgical preparation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric population going under cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2017-09-23 (Actual); Study Completion 2017-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Ueda, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hosptials and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Result] Willschke H, Marhofer P, Bosenberg A, Johnston S, Wanzel O, Sitzwohl C, Kettner S, Kapral S. Epidural catheter placement in children: comparing a novel approach using ultrasound guidance and a standard loss-of-resistance technique. Br J Anaesth. 2006 Aug;97(2):200-7. doi: 10.1093/bja/ael121. Epub 2006 May 23. PMID 16720672
- [Result] Hassan SZ. Caudal anesthesia in infants. Anesth Analg. 1977 Sep-Oct;56(5):686-9. doi: 10.1213/00000539-197709000-00016. PMID 562094
- [Result] Valairucha S, Seefelder C, Houck CS. Thoracic epidural catheters placed by the caudal route in infants: the importance of radiographic confirmation. Paediatr Anaesth. 2002 Jun;12(5):424-8. doi: 10.1046/j.1460-9592.2002.00884.x. PMID 12060329
- [Result] Blanco D, Llamazares J, Rincon R, Ortiz M, Vidal F. Thoracic epidural anesthesia via the lumbar approach in infants and children. Anesthesiology. 1996 Jun;84(6):1312-6. doi: 10.1097/00000542-199606000-00006. PMID 8669671
- [Result] Baidya DK, Pawar DK, Dehran M, Gupta AK. Advancement of epidural catheter from lumbar to thoracic space in children: Comparison between 18G and 23G catheters. J Anaesthesiol Clin Pharmacol. 2012 Jan;28(1):21-7. doi: 10.4103/0970-9185.92429. PMID 22345940
- [Result] Chawathe MS, Jones RM, Gildersleve CD, Harrison SK, Morris SJ, Eickmann C. Detection of epidural catheters with ultrasound in children. Paediatr Anaesth. 2003 Oct;13(8):681-4. doi: 10.1046/j.1460-9592.2003.01151.x. PMID 14535905
- [Result] Tsui BC, Seal R, Koller J. Thoracic epidural catheter placement via the caudal approach in infants by using electrocardiographic guidance. Anesth Analg. 2002 Aug;95(2):326-30, table of contents. doi: 10.1097/00000539-200208000-00016. PMID 12145046
- [Result] Tsui BC, Tarkkila P, Gupta S, Kearney R. Confirmation of caudal needle placement using nerve stimulation. Anesthesiology. 1999 Aug;91(2):374-8. doi: 10.1097/00000542-199908000-00010. PMID 10443599
- [Result] Rapp HJ, Folger A, Grau T. Ultrasound-guided epidural catheter insertion in children. Anesth Analg. 2005 Aug;101(2):333-339. doi: 10.1213/01.ANE.0000156579.11254.D1. PMID 16037140
- [Result] Tsui BC, Berde CB. Caudal analgesia and anesthesia techniques in children. Curr Opin Anaesthesiol. 2005 Jun;18(3):283-8. doi: 10.1097/01.aco.0000169236.91185.5b. PMID 16534352
- [Result] Roberts SA, Galvez I. Ultrasound assessment of caudal catheter position in infants. Paediatr Anaesth. 2005 May;15(5):429-32. doi: 10.1111/j.1460-9592.2004.01512.x. PMID 15828997
- [Result] Owall A, Stahl L, Settergren G. Incidence of sore throat and patient complaints after intraoperative transesophageal echocardiography during cardiac surgery. J Cardiothorac Vasc Anesth. 1992 Feb;6(1):15-6. doi: 10.1016/1053-0770(91)90037-t. PMID 1543845

RESULTS

PARTICIPANT FLOW:
Groups:
- TEE Guided Epidural Catheter Placement: TEE: Epidural catheter will be placed under guidance of transesophageal echography in specific thoracic spinal segment.
Period: Overall Study
Arm/Group | TEE Guided Epidural Catheter Placement
Started | 25
Completed | 20
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- TEE Guided Epidural Cather Placement: TEE: Epidural catheter will be placed under guidance of transesophageal echography in specific thoracic spinal segment.
Arm/Group | TEE Guided Epidural Cather Placement
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Epidural Catheter Placement
Description: The success rate achieved using TEE guidance to thread an epidural catheter to within one targeted thoracic spinal level. Post-operative radiograph will be used to confirm catheter position.
Time Frame: within one day
Measure: Count of Participants; unit: Participants
Arm/Group | TEE Guided Epidural Catheter Placement
Number analyzed (Participants) | 20
Participants
  Successful placement | 17
  Unsuccessful placement | 3

ADVERSE EVENTS:
Time Frame: one day
Arm/Group | TEE Guided Epidural Cather Placement
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-07-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02415998/Prot_SAP_000.pdf
  • Informed Consent Form (2012-07-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02415998/ICF_001.pdf